CLINICAL TRIAL: NCT07383259
Title: Skeletal and Dentoalveolar Effects of Tooth-borne Facemask Versus Skeletal Anchorage Chin-plate Maxillary Protraction in Growing Class III Patients.
Brief Title: Comparison of Maxillary Protraction Using Tooth-borne Facemask Versus Skeletal Anchorage Chin-plate in Class III Growing Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ortoestetic (https://ortoestetic.com) (Unknown)
Responsible Party: Principal Investigator, Concepción Martín Alvaro, Full Professor, Universidad Complutense de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mentoplac_FaceMask
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Skeletal Class III Malocclusion
Keywords: Class III malocclusion; skeletal anchorage; face-mask; Palatal expander; tooth-borne rapid maxillary expander; hybrid skeletal anchorage expander; chin-plate
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: A retrospective non-randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth-Borne Expander with Facemask (FM) (Active Comparator): Bonded acrylic splint-type Hyrax expander with hooks in the maxillary canine region. Expansion activated once daily (0.25 mm). Facemask therapy initiated two weeks after expansion onset with 400 g per side of elastic traction, directed approximately 30° downward relative to the occlusal plane, worn 14-16 hours per day.
  Interventions: Device: Tooth-Borne Expander with Facemask (FM)
- Hybrid Skeletal Anchorage Expander with Chin-Plate (SA) (Experimental): Modified Hybrid Hyrax expander supported by first molars and anchored with miniscrews placed bilaterally in a paramedian position. Expansion activated once daily (0.25 mm). Mandibular chin-plates (bollard-type or single chin-plate depending on eruption stage) were surgically inserted, and Class III elastics delivering 400 g per side were applied following a progressive loading protocol.
  Interventions: Device: Hybrid Skeletal Anchorage Expander with Chin-Plate (SA)

INTERVENTIONS:
Device: Tooth-Borne Expander with Facemask (FM) — Bonded acrylic splint-type Hyrax expander with hooks in the maxillary canine region. Expansion activated once daily (0.25 mm). Facemask therapy initiated two weeks after expansion onset with 400 g per side of elastic traction, directed approximately 30° downward relative to the occlusal plane, worn 14-16 hours per day.
  Arms: Tooth-Borne Expander with Facemask (FM)
Device: Hybrid Skeletal Anchorage Expander with Chin-Plate (SA) — Modified Hybrid Hyrax expander supported by first molars and anchored with miniscrews placed bilaterally in a paramedian position. Expansion activated once daily (0.25 mm). Mandibular chin-plates (bollard-type or single chin-plate depending on eruption stage) were surgically inserted, and Class III elastics delivering 400 g per side were applied following a progressive loading protocol.
  Arms: Hybrid Skeletal Anchorage Expander with Chin-Plate (SA)

SUMMARY:
This retrospective non-randomized controlled clinical trial aimed to compare the skeletal and dentoalveolar effects of two orthopedic treatment protocols for skeletal Class III malocclusion in growing patients: a conventional tooth-borne rapid maxillary expansion combined with facemask therapy, and a hybrid skeletal anchorage expander combined with chin-plate traction. Lateral cephalometric changes before and after maxillary protraction were analyzed to assess sagittal skeletal correction and dentoalveolar effects.

DETAILED DESCRIPTION:
Skeletal Class III malocclusion is frequently associated with maxillary growth deficiency and presents significant functional and esthetic challenges. Conventional treatment using rapid maxillary expansion combined with facemask therapy is effective but limited by patient compliance and undesirable dentoalveolar effects. The introduction of skeletal anchorage devices allows the application of orthopedic forces with reduced dental compensation and extended effectiveness beyond early growth stages.

This study retrospectively evaluated growing patients (CVS1-CVS3) treated with either a tooth-borne expander and facemask or a hybrid skeletal anchorage expander combined with chin-plate traction. Cephalometric variables were measured before treatment (T0) and after completion of maxillary protraction (T1) to compare skeletal and dentoalveolar changes between protocols.

ELIGIBILITY:
Inclusion Criteria

* Growing patients (CVS1-CVS3)
* Patent midpalatal suture (stages A-C)
* Skeletal Class III malocclusion (ANB < 0°, Wits < -2 mm)
* Presence of anterior crossbite or edge-to-edge incisal relationship Exclusion Criteria
* Severe craniofacial asymmetry
* Evidence of active condylar growth
* Previous orthodontic treatment
* Craniofacial malformations or syndromes
* Systemic diseases or medications affecting growth or bone metabolism

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in sagittal skeletal relationship | From baseline (T0) through study completion, an average of 1 year (T1)
  Changes in the cephalometric angles SNA, ANB, and Wits appraisal measured on lateral cephalograms between T0 and T1

SECONDARY OUTCOMES:
Cephalometric vertical skeletal changes | From baseline (T0) through study completion, an average of 1 year (T1)
  o Cephalometric vertical measurements from T0 to T1, using a customized cephalometric analysis based on Steiner, Tweed, and McNamara references: Mandibular plane to SN (Sella-Nasion) angle, ANS (Anterior Nasal Spine)-PNS (Posterior Nasal Spine) to Mandibular plane angle, and ANS-PNS to SN angle
Cephalometric dentoalveolar changes | From baseline (T0) through study completion, an average of 1 year (T1)
  o Upper and lower incisor inclination changes from T0 to T1 using a customized cephalometric analysis based on Steiner, Tweed, and McNamara references: U_SN (Upper incisor to Sella-Nasion)and IMPA (Lower Incisor Mandibular Plane Angle)
Treatment duration | From baseline (T0) through study completion, an average of 1 year (T1)
  o Time elapsed between T0 and T1

IPD SHARING:
Plan to Share IPD: Undecided
Upon request